CLINICAL TRIAL: NCT00512889
Title: A Pilot Study of the Adoptive Transfer of MART1/Melan-A CTL for Malignant Melanoma
Brief Title: Adoptive Transfer of MART1/Melan-A CTL for Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Marcus O. Butler, MD, Instructor, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-250
Record Dates: First submitted 2007-08-03; First posted 2007-08-08 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Melanoma (Skin)
Keywords: CTL; MART-1; Melan-A; artificial APC; melanoma; metastatic melanoma; adoptive immunotherapy; adoptive cell transfer; immunotherapy
MeSH Terms: conditions — Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Different dose of CTL
  Interventions: Biological: therapeutic autologous lymphocytes; Genetic: Use of an artificial antigen presenting cell (aAPC) to generate CTL
- Cohort 2 (Experimental): Different dose of CTL
  Interventions: Biological: therapeutic autologous lymphocytes; Genetic: Use of an artificial antigen presenting cell (aAPC) to generate CTL
- Cohort 3 (Experimental): Combination of CTL with GMCSF +/- radiation
  Interventions: Biological: therapeutic autologous lymphocytes; Genetic: Use of an artificial antigen presenting cell (aAPC) to generate CTL; Drug: GM-CSF; Radiation: Irradiation of cutaneous tumor lesion

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes — Autologous CTL generated from peripheral blood following culture with MART1/Melan-A peptide pulsed aAPC.
Genetic: Use of an artificial antigen presenting cell (aAPC) to generate CTL — A genetically modified artificial antigen presenting cell (aAPC) is used in the generation of anti-tumor CTL.
Drug: GM-CSF — GM-CSF will be used as an immune activator and combined with the infusion of MART1/Melan-A specific CTL.
  Arms: Cohort 3
Radiation: Irradiation of cutaneous tumor lesion — Irradiation of cutaneous melanoma lesion will be combined with the infusion of MART1/Melan-A specific CTL.
  Arms: Cohort 3

SUMMARY:
RATIONALE: Cytotoxic T lymphocytes (CTL) are cells of the immune system that can fight infections and cancer. These CTL can be manipulated in the laboratory so that they can target an individual's cancer.

PURPOSE: This early phase trial is studying the feasibility and side effects of intravenous infusions of CTL generated in the laboratory. To produce the CTL, the study participant's own immune cells are collected by a procedure called a leukapheresis. The cells then undergo laboratory processing for three weeks. Part of this processing includes mixing the patients immune cells with a new kind of cell that has some extra genes added to it. These extra genes are to "teach" the participant's own immune cells to become anti-tumor CTL that can attack the melanoma.

DETAILED DESCRIPTION:
DETAILED OUTLINE: This is an early phase pilot/feasibility trial.

Study subjects will be sequentially accrued to three cohorts. Cohorts 1 and 2 will evaluate the safety and feasibility of infusing two different doses of CTL.

* Participants in all cohorts will undergo two CTL infusions 5 weeks apart.
* Procedures performed during the trial will include physical examinations, laboratory tests, delayed hypersensitivity testing, and skin biopsies.
* Between 5 and 8 days after the first CTL infusion, a biopsy or excision of a melanoma lesion may be performed.
* Three leukapheresis procedures will be performed: two to collect peripheral blood for CTL production and one for research purposes at the end of the clinical trial.
* Radiology tests (including CT scans) will be performed prior to infusion and about 4-5 weeks after the second CTL infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic melanoma: Either unresectable Stage III or any Stage IV
* ECOG of 0 or 1
* HLA-A*0201 haplotype
* Baseline tumor biopsy MART1/Melan-A expression present (in >10% of tumor cells)
* Patient provides consent for all required biopsies
* Adequate intravenous access for leukapheresis
* Absolute lymphocyte count >500/ul at least once within 30 days of leukapheresis
* Life expectancy greater than 4 months in the opinion of the study clinician
* Negative pregnancy test

Exclusion Criteria:

* Administration of systemic corticosteroids within 28 days of planned leukapheresis
* Administration of cytotoxic chemotherapy or anti-tumor immunotherapy within 28 days of planned leukapheresis
* Administration of radiotherapy within 28 days of planned leukapheresis with the exception of subjects accrued to Cohort 3
* Active autoimmunity requiring systemic immunosuppressive therapy
* HIV infection
* Previous enrollment on this protocol and infusion of MART1/Melan-A CTL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-08; Primary Completion 2011-02 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Define the feasibility of generating large doses of MART1/Melan-A specific CTL following leukapheresis in this patient population | 2 years
Describe the toxicity of two dose levels of adoptively transferred MART1/Melan-A specific CTL lines | 2 years
Define the feasibility of combining the infusion of MART1/Melan-A specific CTL with the administration of GM-CSF +/- radiotherapy | 2 years
Describe the toxicity of combining the infusion of MART1/Melan-A specific CTL with the administration of GM-CSF +/- radiotherapy | 2 years

SECONDARY OUTCOMES:
Evaluate function, phenotype, and trafficking of infused CTL. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Butler, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Result] Butler MO, Friedlander P, Milstein MI, Mooney MM, Metzler G, Murray AP, Tanaka M, Berezovskaya A, Imataki O, Drury L, Brennan L, Flavin M, Neuberg D, Stevenson K, Lawrence D, Hodi FS, Velazquez EF, Jaklitsch MT, Russell SE, Mihm M, Nadler LM, Hirano N. Establishment of antitumor memory in humans using in vitro-educated CD8+ T cells. Sci Transl Med. 2011 Apr 27;3(80):80ra34. doi: 10.1126/scitranslmed.3002207. PMID 21525398